CLINICAL TRIAL: NCT01741870
Title: The Effectiveness of a Need-based Nutritional Intervention Strategy to Improve the Nutritional Status of Elderly Nursing Home Residents
Brief Title: A Need-based Nutritional Intervention in Nursing Home Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: tsai1943
Record Dates: First submitted 2012-11-29; First posted 2012-12-05 (Estimated); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Malnutrition
Keywords: Nutritional supplement; Nutritional status; Physical functional activity; Nursing home elderly
MeSH Terms: conditions — Malnutrition | interventions — Dietary Supplements; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): No intervention was given. All subjects received routine care
  Interventions: Other: Treatment as usual
- Received nutrition supplement as needed (Active Comparator): Subjects in this group received 50 g/day soy protein-based nutritional supplement (containing 9.5 g protein, 250 kcal energy and all essential micro-nutrients) whenever subjects BMI is below 24 and MNA score also below 24.
  Interventions: Dietary Supplement: Nutritional supplement; Other: Treatment as usual

INTERVENTIONS:
Dietary Supplement: Nutritional supplement — Subjects will receive 50 g/day of a soy protein-based nutritional supplement containing 9.5 g protein, 250 kcal energy and all essential micronutrients
  Arms: Received nutrition supplement as needed
Other: Treatment as usual — routine care

SUMMARY:
To examine the effectiveness of a "need-based nutritional intervention" strategy in improving the nutritional and physical functional status of nursing home elderly.

DETAILED DESCRIPTION:
Ninety-two nursing home residents aged 65 years or older and BMI <25 were randomly assigned to the intervention or control groups. Subjects in the treatment group received a soy-protein-based nutritional supplement, if his/her BMI was <24kg/m2 and nutritional score was <24 according to the Mini Nutritional Assessment. The supplementation would be suspended if both conditions were not met. At baseline and every 4 weeks up to 24 weeks, thereafter, all subjects were measured for anthropometric parameters. At baseline, 12 weeks and 24 weeks subjects were measured for blood biochemical indicators, handgrip strength and Barthel's index.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 65 years of age
2. BMI ≤ 25 (kg/m2)
3. ≥1 month of residency
4. Able to self-feed or receive oral-feeding
5. Non-bed-ridden
6. Cognitively able to answer the questionnaire

Exclusion Criteria:

1.Hospitalized or having acute infection/diseases

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 92 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Assessment of nutritional status with the Mini nutritional Assessment (MNA) | Baseline and every 4 weeks, up to 24 weeks
  Change from baseline in MNA score at 4, 8, 12, 16, 20 and 24 weeks

SECONDARY OUTCOMES:
Biochemical indicators | Baseline, 12, and 24 weeks
  Change from baseline in serum albumin and cholesterol concentrations, and hemoglobin, hematocrit and lymphocyte count status at 12, and 24 weeks.

OTHER OUTCOMES:
Physical functional status | Baseline, 12 and 24 weeks
  Change from baseline in Barthel's index and handgrip strength at 12 and 24 weeks
Hospital admissions | Baseline, and 24 weeks
  Frequency of outpatient visits, emergency visits and hospital admission (length of stay) during the study

CONTACTS AND LOCATIONS:
Overall Officials: Alan C Tsai, PhD, Principal Investigator — Professor, Dept. of Healthcare Adm., Asia University, 500 liufeng Road, Wufeng, Taichung, Taiwan 41354
Locations (1):
- Asia University, Taichung, Taiwan

REFERENCES:
- [Background] Weatherall M. Protein-energy oral supplementation in malnourished nursing-home residents. Age Ageing. 2001 Jan;30(1):85. doi: 10.1093/ageing/30.1.85. No abstract available. PMID 11322680
- [Derived] Lee LC, Tsai AC, Wang JY, Hurng BS, Hsu HC, Tsai HJ. Need-based intervention is an effective strategy for improving the nutritional status of older people living in a nursing home: a randomized controlled trial. Int J Nurs Stud. 2013 Dec;50(12):1580-8. doi: 10.1016/j.ijnurstu.2013.04.004. Epub 2013 May 3. PMID 23648392